CLINICAL TRIAL: NCT00705601
Title: Refinement Of Patient Reported Outcomes Instruments In Subjects With Insomnia Characterized By Nonrestorative Sleep
Brief Title: Nonrestorative Sleep RSQ (Restorative Sleep Questionnaire) Development-- Methodology Study
Status: Terminated | Type: Observational
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A9001380
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Nonrestorative Sleep
Keywords: Nonrestorative Sleep, Restorative Sleep Questionnaire Refinement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: PSG

INTERVENTIONS:
Procedure: PSG — PSG (polysomnography) for adaptation night, day 2 evening, and day 3 evening--used to identify suitable Nonrestorative Sleep candidates to participate in focus groups.

SUMMARY:
To begin to refine development of the RSQ (Restorative Sleep Questionnaire) measure in subjects with NRS (Nonrestorative Sleep) by generating item content pertaining to morning refreshment and uncovering problems in instrument administration in subjects with nonrestorative sleep

DETAILED DESCRIPTION:
Study was terminated on January 20, 2009 due to portfolio decision by Pfizer to discontinue further investigation of PD200390 for non-restorative sleep. The decision was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who self report nonrestorative sleep but no problems either getting to sleep or staying asleep
* Complaints of significant distress or impairment in social, occupational, or other important areas of functioning during daytime for at least 3 nights per week
* Self reports sWASO (Wake after sleep onset) for <45 minutes for past 3 months, self reports LPS (latency to persistent sleep onset ) for <20 minutes for past 3 months (then neither PSG (polysomnography) screening night showing WASO >45min, or LPS > 20 minutes)
* Customary bedtime betw. 9 pm and midnight and rise between 4 and 9 AM

Exclusion Criteria:

* Psychiatric disease or disorder as determined by current administration of the MINI (Mini International Neuropsychiatric Interview)
* History or presence of any breathing-related sleep disorder, narcolepsy, or any other dyssomnias or any parasomnia, or restless legs syndrome MAP > 0.5 at screening
* History or presence of any medical or neurological condition that could interfere with sleep (chronic pain, Restless leg, etc)
* Current use of meds wth known psychotropic effects or known or suspected effects on sleep
* Alcohol or substance abuse (unless in remission for at least a year
* Excessive caffeine use (or any use after 6 pm for at least 3 months
* Regular napping or any naps after 6 pm
* Excessive cigarette or cigar smoking over the last 3 months
* no participation in an investigational new drug study within 30 days of screening, and no previous participation in a study of PD200390
* No night or rotating shift work

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Once subjects identified, a series of focus group sessions will be held to identify concepts, themes and items relevant to Nonrestorative Sleep. | monthly
To begin to refine the development of the RSQ measure in subjects with Nonrestorative Sleep by generating item content pertaining to morning refreshment and uncovering problems in instrument administration in subjects with nonrestorative sleep. | nightly
Identification of subjects with insomnia characterized by Nonrestorative Sleep only [assessed via LPS (latency to persistent sleep onset) and WASO (Wake after sleep onset) as determined by PSG (polysomnography)]. | nightly

SECONDARY OUTCOMES:
Subjective measures include MAF (multidimensional assessment of fatigue), Sheehan Disability Scale, SF36v2, Endicott Work productivity scale (EWPS) Global impression of severity (CGIS) and the Profile of mood states. | nightly
Secondary assessments to characterize the functional impact of insomnia including Nonrestorative Sleep include additional PSG (polysomnography) variables. | nightly
After phase IIa of this study, a questionaire to be designed - Participants to be debriefed, and interviewed to assess the content validity of the questionnaire. | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (11):
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Columbus, Ohio
- Canada (2):
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Drake CL, Hays RD, Morlock R, Wang F, Shikiar R, Frank L, Downey R, Roth T. Development and evaluation of a measure to assess restorative sleep. J Clin Sleep Med. 2014 Jul 15;10(7):733-41, 741A-741E. doi: 10.5664/jcsm.3860. PMID 25024650
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001380&StudyName=Nonrestorative%20Sleep%20RSQ%20%28Restorative%20Sleep%20Questionnaire%29%20Development--%20Methodology%20Study